CLINICAL TRIAL: NCT02744937
Title: To Investigate Post-procedure Hemorrhage and Cardiovascular Events in Taiwanese Patients Who Continue or Discontinue Low-Dose Aspirin Before Transrectal Prostate Biopsy: a Prospective Randomized Trial
Brief Title: Continuing Low Dose Aspirin Before Prostate Biopsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, V.S., National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201601033MINC
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Complication
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): continuing LDA
  Interventions: Drug: Aspirin
- B (No Intervention): discontinuing LDA

INTERVENTIONS:
Drug: Aspirin — aspirin is continued by its regular dosing
  Arms: A

SUMMARY:
Objectives: To determine whether TRUS-guided prostate biopsy performed in patients continuing low-dose aspirin (LDA) is associated with a greater incidence, duration, and severity of bleeding complications.

Eligibility: Men over 40-year-old with an elevated serum prostate-speciﬁc antigen level and/or abnormal digital rectal examination ﬁndings are candidates for PB.

Design of trial Prospective Randomized Trial Study treatment: Continuing low-Dose aspirin before transrectal prostate biopsy Primary endpoint: The incidence, duration, and severity of bleeding complications Statistical analysis and sample size estimation: Fisher's exact test or chi-square test will be used to explore the differences between two groups for categorical variables, and Student t-test will be used for continuous variables. Under the assumption of a difference of 25% of bleeding complications in each group, with α=0.05 and power=0.80, 60 subject are needed in each arm. Assuming the drop-out rate to be 20%, the targeted recruit number is 150 in total.

DETAILED DESCRIPTION:
Transrectal ultrasound (TRUS)-guided prostate biopsy (PB) is currently the standard for diagnosing prostate cancer and is one of the most commonly performed urologic procedures.

The complications that can occur after this procedure have been extensively described previously. Bleeding complications, namely hematuria, rectal bleeding, and hematospermia, are the most frequent, with a reported incidence of 20% to 70%, but they are almost exclusively self-limiting and of mild to moderate severity.

There is an increasing number of patients who require PB and antiplatelet medication simultaneously. This is because more middle-age and elderly patients are receiving long-term antithrombotic therapy mainly for prevention of cardiovascular events, and these patients form the majority of those at risk of prostate cancer. As with other surgical interventions, aspirin is typically discontinued 7 to 10 days before PB. However, discontinuing aspirin might increase the risk of cardiovascular events, while continuing aspirin before PB might not necessarily increase severe bleeding complications. Several studies have found no increase in bleeding complications in patients continuing low-dose aspirin. However, most of the studies were retrospective, and only one was randomized. Moreover, there has been no prospective randomized trial in East Asian patients, who have a lower risk of thrombosis and increased risk of bleeding during antithrombotic treatment for acute coronary syndrome than do white patients.

The aim of the present randomized study was to determine whether TRUS-guided PB performed in patients continuing low-dose aspirin (LDA) is associated with a greater incidence, duration, and severity of bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are use of LDA (100 mg once daily) for primary prevention of cardiovascular disease and not at a high risk of cardiovascular event. The definition of high risk includes #1-7 of the following exclusion criteria or unsuitable conditions by clinical judgement.

Exclusion Criteria:

1. Angina in the past 3 months
2. Exertional dyspnea on walking or climbing stairs for one floor
3. Stroke in the past 6 months
4. Coronary catheterization in the past 6 months
5. Left main disease or 3-vessel disease
6. Prior coronary arterial bypass graft surgery
7. Use of dual (or more) antiplatelet agents
8. Coagulopathy or diseases with bleeding tendency
9. Hemorrhoid, anal or rectal diseases
10. History of urinary stone or tumor

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Compications | 3 weeks
  To determine whether the incidence, duration, and severity of bleeding complications after transrectal prostate biopsy (PB) in patients not discontinuing low-dose aspirin (LDA) are greater than in those discontinuing it.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maan Z, Cutting CW, Patel U, Kerry S, Pietrzak P, Perry MJ, Kirby RS. Morbidity of transrectal ultrasonography-guided prostate biopsies in patients after the continued use of low-dose aspirin. BJU Int. 2003 Jun;91(9):798-800. doi: 10.1046/j.1464-410x.2003.04238.x. PMID 12780835
- [Result] Berger AP, Gozzi C, Steiner H, Frauscher F, Varkarakis J, Rogatsch H, Bartsch G, Horninger W. Complication rate of transrectal ultrasound guided prostate biopsy: a comparison among 3 protocols with 6, 10 and 15 cores. J Urol. 2004 Apr;171(4):1478-80; discussion 1480-1. doi: 10.1097/01.ju.0000116449.01186.f7. PMID 15017202
- [Result] Ihezue CU, Smart J, Dewbury KC, Mehta R, Burgess L. Biopsy of the prostate guided by transrectal ultrasound: relation between warfarin use and incidence of bleeding complications. Clin Radiol. 2005 Apr;60(4):459-63; discussion 457-8. doi: 10.1016/j.crad.2004.10.014. PMID 15767103
- [Result] Chiang IN, Chang SJ, Pu YS, Huang KH, Yu HJ, Huang CY. Major complications and associated risk factors of transrectal ultrasound guided prostate needle biopsy: a retrospective study of 1875 cases in taiwan. J Formos Med Assoc. 2007 Nov;106(11):929-34. doi: 10.1016/S0929-6646(08)60063-7. PMID 18063514
- [Result] Ehrlich Y, Yossepowitch O, Margel D, Lask D, Livne PM, Baniel J. Early initiation of aspirin after prostate and transurethral bladder surgeries is not associated with increased incidence of postoperative bleeding: a prospective, randomized trial. J Urol. 2007 Aug;178(2):524-8; discussion 528. doi: 10.1016/j.juro.2007.03.134. Epub 2007 Jun 14. PMID 17570430
- [Result] Giannarini G, Mogorovich A, Valent F, Morelli G, De Maria M, Manassero F, Barbone F, Selli C. Continuing or discontinuing low-dose aspirin before transrectal prostate biopsy: results of a prospective randomized trial. Urology. 2007 Sep;70(3):501-5. doi: 10.1016/j.urology.2007.04.016. Epub 2007 Aug 3. PMID 17688919
- [Result] Ecke TH, Gunia S, Bartel P, Hallmann S, Koch S, Ruttloff J. Complications and risk factors of transrectal ultrasound guided needle biopsies of the prostate evaluated by questionnaire. Urol Oncol. 2008 Sep-Oct;26(5):474-8. doi: 10.1016/j.urolonc.2007.12.003. Epub 2008 Mar 4. PMID 18367116
- [Result] Halliwell OT, Yadegafar G, Lane C, Dewbury KC. Transrectal ultrasound-guided biopsy of the prostate: aspirin increases the incidence of minor bleeding complications. Clin Radiol. 2008 May;63(5):557-61. doi: 10.1016/j.crad.2007.09.014. Epub 2008 Jan 11. PMID 18374720
- [Result] Carmignani L, Picozzi S, Bozzini G, Negri E, Ricci C, Gaeta M, Pavesi M. Transrectal ultrasound-guided prostate biopsies in patients taking aspirin for cardiovascular disease: A meta-analysis. Transfus Apher Sci. 2011 Dec;45(3):275-80. doi: 10.1016/j.transci.2011.10.008. Epub 2011 Oct 24. PMID 22030310
- [Result] Chowdhury R, Abbas A, Idriz S, Hoy A, Rutherford EE, Smart JM. Should warfarin or aspirin be stopped prior to prostate biopsy? An analysis of bleeding complications related to increasing sample number regimes. Clin Radiol. 2012 Dec;67(12):e64-70. doi: 10.1016/j.crad.2012.08.005. Epub 2012 Sep 7. PMID 22959852
- [Result] Raheem OA, Casey RG, Galvin DJ, Manecksha RP, Varadaraj H, McDermott T, Grainger R, Lynch TH. Discontinuation of anticoagulant or antiplatelet therapy for transrectal ultrasound-guided prostate biopsies: a single-center experience. Korean J Urol. 2012 Apr;53(4):234-9. doi: 10.4111/kju.2012.53.4.234. Epub 2012 Apr 18. PMID 22536465
- [Result] Wang J, Zhang C, Tan G, Chen W, Yang B, Tan D. Risk of bleeding complications after preoperative antiplatelet withdrawal versus continuing antiplatelet drugs during transurethral resection of the prostate and prostate puncture biopsy: a systematic review and meta-analysis. Urol Int. 2012;89(4):433-8. doi: 10.1159/000343733. Epub 2012 Nov 13. PMID 23154789
- [Result] Culkin DJ, Exaire EJ, Green D, Soloway MS, Gross AJ, Desai MR, White JR, Lightner DJ. Anticoagulation and antiplatelet therapy in urological practice: ICUD/AUA review paper. J Urol. 2014 Oct;192(4):1026-34. doi: 10.1016/j.juro.2014.04.103. Epub 2014 May 21. PMID 24859439